CLINICAL TRIAL: NCT01134744
Title: Study of Accuracy of Clinical Examination for Chest Trauma
Brief Title: Evaluating Validity of Clinical Criteria for Requesting Chest X-Rays in Trauma Patients
Status: Completed | Type: Observational
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy, Associate Professor of Medical Education, Isfahan University of Medical Sciences
Other Study IDs: ASD-1213-3
Record Dates: First submitted 2010-05-27; First posted 2010-06-02 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2006-10

CONDITIONS: Chest Trauma
Keywords: CXray
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chest trauma: chest x-ray applied for patients with chest trauma and the manifestations compared with clinical examination

SUMMARY:
The purpose of this study is to identify the clinical criteria for requesting a chest x-ray in a patient with blunt trauma and its findings such as clinical signs with a high sensitivity could be used in a larger study to codify the final criteria.

DETAILED DESCRIPTION:
At present, a Chest x-ray is obtained from all trauma patients having suspicion to chest trauma. The indications for such radiographs are not well defined. This results in a large number of unnecessary chest radiographs being obtained. Our goal was to identify the clinical criteria for requesting a chest x-ray in a patient with blunt trauma and its findings such as clinical signs with a high sensitivity could be used in a larger study to codify the final criteria.

ELIGIBILITY:
Inclusion Criteria:

* Every patient with blunt trauma to chest

Exclusion Criteria:

* nothing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three hundred and eighty six
Sampling Method: Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
chest pain | 5 min after admision time
  for Assessing the accuaracy of this outcome we evaluated this one with chest x-ray manifestation

SECONDARY OUTCOMES:
tachypnea | 5 min after admision time
  for Assessing the accuaracy of this outcome we evaluated this one with chest x-ray manifestation
abrasion | 5 min after admision time
  for Assessing the accuaracy of this outcome we evaluated this one with chest x-ray manifestation
crepitation | 5 min after admision time
  for Assessing the accuaracy of this outcome we evaluated this one with chest x-ray manifestation

CONTACTS AND LOCATIONS:
Overall Officials: hamidreza shemshaki, MD, Study Chair — MD,research comittee
Locations (2):
- Iran (2):
  - Al-zahra university hospital, Isfahan
  - Emamkhomeini University Hospital, Tehran